CLINICAL TRIAL: NCT04684056
Title: Laboratory Assessment of the Anticoagulant Activity of Direct Oral Anticoagulants in Peri-operative Catheter Ablation for Patient With Atrial Fibrillation
Brief Title: Laboratory Assessment of the Concentration of Direct Oral Anticoagulants in Patients With Atrial Fibrillation
Acronym: LOAF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Collaborators: Wuhan Asia General Hospital (http://wagh.com.cn) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-YXKY-B010
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Oral Anticoagulant; Atrial Fibrillation; Pharmacokinetics and Pharmacodynamics
Keywords: Direct oral anticoagulants; pharmacokinetics and pharmacodynamics; Atrial Fibrillation; Rivaroxaban; Dabigatran; Edoxaban; Anti-FXa assays; Dilute thrombin time; Liquid-chromatography tandem mass spectrometry
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Riva-control group: Routine concentration of Rivaroxaban (Peak)
- Riva-High group: High concentration of Rivaroxaban (Peak)
- Riva-Low group: low concentration of Rivaroxaban (Peak)
- Dabi-control group: Routine concentration of Dabigatran(Peak)
- Dabi-High group: High concentration of Dabigatran(Peak)
- Dabi-low group: low concentration of Dabigatran(Peak)
- Edo-control group: Routine concentration of Edoxaban(Peak)
- Edo-high group: High concentration of Edoxaban(Peak)
- Edo-low group: low concentration of Edoxaban(Peak)

SUMMARY:
The incidence of thromboembolic and bleeding event associated with catheter ablation for atrial fibrillation(CAAF) varies from 0.9% to 5% during peri-operative period. Direct oral anticoagulants (DOAC) (such as Rivaroxaban, Dabigatran and Edoxaban) are gradually applied in clinical practice to prevent thrombosis events in patients with AF, but studies have shown that DOAC are also affected by surgery, an invasive procedure, sub-therapeutic, food, renal function and age. However, the pharmacokinetic and pharmacodynamic of DOAC during the peri-operative period of CAAF were lacking in China. The purpose of this study was to evaluate the pharmacokinetics and pharmacokinetics of DOAC in patients with peri-operative atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Non-valvular atrial fibrillation(NVAF) undergoing catheter ablation
* Direct oral anticoagulants (Rivaroxaban, Edoxaban or Dabigatran)are administered peri-operatively during catheter ablation.

Exclusion Criteria:

* Patients who have taken direct oral anticoagulants or warfarin before admission.
* Cross-replacement of oral anticoagulants, such as taking dabigatran before surgery and replacing Rivaroxaban after surgery.
* Abnormal coagulation tests (prothrombin time, partial thrombin time, thrombin time, antithrombin activity).
* Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Catheter ablation was performed under general anesthesia in patients with NVAF. Direct oral anticoagulants (Rivaroxaban, Edoxaban or Dabigatran )were administered peri-operatively to prevent thrombotic events.
Sampling Method: Probability Sample
Enrollment: 1864 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of thromboembolic | Ninety days after catheter ablation
  Ischemic stroke, Deep vein thrombosis (DVT) or arterial thrombosis of any location after taking DOAC
Bleeding Incidence | Ninety days after catheter ablation
  Any bleeding, Especially gastrointestinal hemorrhage or hemoglobin drop is greater than 20g/L after taking DOAC

SECONDARY OUTCOMES:
Death from any cause | Ninety days after catheter ablation